CLINICAL TRIAL: NCT01289015
Title: A Phase 3 Double-Blind, Randomized, Placebo-Controlled,Multicenter, Parallel Group Evaluation of the Efficacy and Safety of NAFT-600 in Subjects With Tinea Pedis
Brief Title: Efficacy and Safety of NAFT-600 in Subjects With Tinea Pedis
Acronym: NAFT-600
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merz North America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MRZ 90200/3015/1
Record Dates: First submitted 2011-01-28; First posted 2011-02-03 (Estimated); Results first posted 2013-09-26 (Estimated); Last update posted 2013-09-26 (Estimated); Status verified 2013-07

CONDITIONS: Tinea Pedis
Keywords: fungal infection; athlete foot
MeSH Terms: conditions — Tinea Pedis; Mycoses | interventions — naftifine; Gels

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NAFT-600 ( naftin 2 % gel) (Experimental)
  Interventions: Drug: NAFT-600 ( naftin 2 % gel )
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NAFT-600 ( naftin 2 % gel ) — Topical; applied once daily for two weeks
  Arms: NAFT-600 ( naftin 2 % gel)
Drug: Placebo — Topical; applied once daily for two weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of NAFT-600, applied once daily for 2 weeks, when compared to placebo for 2 weeks in the treatment of subjects with tinea pedis.

ELIGIBILITY:
Inclusion Criteria:

* Males or non-pregnant females, ≥12 years of age, of any race or sex. Females of child-bearing potential must have a negative urine pregnancy test.
* Presence of interdigital only or both interdigital and moccasin types of tinea pedis on one or both feet characterized by clinical evidence of a tinea infection (at least moderate erythema, moderate scaling and mild pruritus) based on signs and symptoms in the affected area(s)).

Exclusion Criteria:

* Subjects with life-threatening condition (ex. autoimmune deficiency syndrome, cancer,unstable angina or myocardial infarction) within the last 6 months.
* Subjects with abnormal findings - physical or laboratory - that are considered by the investigator to be clinically important and indicative of conditions that might complicate interpretation of study results.
* Subjects with a known hypersensitivity to study drugs or their components.
* Subjects who have a recent history or who are currently known to abuse alcohol or drugs.
* Uncontrolled diabetes mellitus.
* Hemodialysis or chronic ambulatory peritoneal dialysis therapy.
* Current diagnosis of immunocompromising conditions.
* Foot psoriasis, corns and/or callus involving any web spaces, atopic or contact dermatitis.
* Severe dermatophytoses, onychomycosis (on the evaluated foot), mucocutaneous candidiasis or bacterial skin infection.
* Extremely severe tinea pedis (incapacitating).
* Female subject who is pregnant or lactating, who is not using or does not agree to use an acceptable form of contraception during the study, or who intends to become pregnant during the study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 855 (Actual)
Dates: Start 2011-02; Primary Completion 2011-11 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Parish, MD, Principal Investigator — Paddington Testing Co., Inc.
Locations (23):
- United States (22):
  - Associated Foot & Ankle Specialists, LLC, Phoenix, Arizona
  - Skin Surgery Medical Group, Inc., San Diego, California
  - UCSF Dermatology Research, San Francisco, California
  - The Savin Center, PC, New Haven, Connecticut
  - Avail Clinical Research, DeLand, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - International Dermatology Research, Inc., Miami, Florida
  - Miami Dermatology Research Institute, LLC, North Miami Beach, Florida
  - Radiant Research, Inc., Pinellas Park, Florida
  - Northwest Clinical Trials, Boise, Idaho
  - Physician Skin Care, Louisville, Kentucky
  - Michigan Center for Skin Care Research, Clinton Township, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Skin Search of Rochester, Inc., Rochester, New York
  - Crescent Medical Research, Salisbury, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Paddington Testing Co., Inc., Philadelphia, Pennsylvania
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - DermResearch, Inc., Austin, Texas
  - The Center for Skin Research, Houston, Texas
  - Endeavor Clinical Trials, PA, San Antonio, Texas
- Advanced Medical Concepts, PSC, Cidra, PR, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Groups:
- NAFT-600: NAFT-600 : Topical; applied once daily for two weeks
- Placebo: Placebo : Topical; applied once daily for two weeks
Period: Overall Study
Arm/Group | NAFT-600 | Placebo
Started | 571 | 284
Completed | 472 | 230
Not Completed | 99 | 54
Not completed — Protocol Violation | 12 | 9
Not completed — Adverse Event | 3 | 0
Not completed — Lost to Follow-up | 33 | 17
Not completed — Withdrawal by Subject | 17 | 8
Not completed — Disease progression | 1 | 0
Not completed — Negative baseline culture and others | 33 | 20

BASELINE CHARACTERISTICS:
Population: The Safety Evaluation Set (SES) which is the population of subjects who received at least one dose of study medication was used.
Groups:
- Total: Total of all reporting groups
Arm/Group | NAFT-600 | Placebo | Total
Number analyzed (Participants) | 571 | 284 | 855
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 2 | 7
  Between 18 and 65 years | 524 | 255 | 779
  >=65 years | 42 | 27 | 69
Age Continuous [Mean (Standard Deviation); unit: years] | 45.3 (13.3) | 46.4 (14.3) | 45.7 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 416 | 221 | 637
  Male | 155 | 63 | 218
Region of Enrollment [Number; unit: participants]
  United States | 545 | 271 | 816
  Puerto Rico | 26 | 13 | 39

OUTCOME MEASURES:

1. Primary Outcome: Complete Cure of Interdigital Tinea Pedis
Description: The primary efficacy comparison between NAFT-600 gel and placebo will be based on the percentage of subjects at Week 6 with complete cure of interdigital tinea pedis.
  Complete cure is defined as negative mycology results (dermatophyte culture and KOH) and the absence of erythema, scaling, and pruritus.
Time Frame: Visit 4/ Week 6
Population: Full Analysis Set (FAS) defined as the subset of all subjects in the Safety Evaluation Set (SES) with a positive mycology culture at baseline and for whom the primary efficacy variable is available. This was a modified intent to treat principle because culture results were not available before the start of treatment.
Measure: Number; unit: percentage of subjects
Arm/Group | NAFT-600 | Placebo
Number analyzed (Participants) | 382 | 179
percentage of subjects | 16.8 | 1.7
Statistical Analysis 1: Comparison: NAFT-600 vs Placebo; In order to compare complete cure rate in the NAFT-600 group with that of the placebo group, the following one-sided hypothesis test was carried out: H0 (null): p1<=p0 versus Ha (alternate): p1>p0, where p0 and p1 are the proportions of subjects with complete cure in the proportions of subjects with complete cure in the placebo and NAFT-600 treatment groups respectively; Test type: Superiority or Other; p < 0.025, Cochran-Mantel-Haenszel; The CMH test statistic after stratification was used to compare subjects with complete cure between NAFT-600 and placebo; p-value = 0.001

2. Secondary Outcome: Effective Treatment and Mycological Cure of Interdigital Tinea Pedis at Week 6
Description: Effective treatment of interdigital tinea pedis which is defined as negative KOH and negative dermatophyte culture and erythema, scaling, and pruritus scores of 0 or 1 (corresponding to absent and mild respectively).
  Mycological cure of interdigital tinea pedis which is defined as negative KOH and negative dermatophyte culture.
Time Frame: Visit 4/ Week 6.
Population: Full Analysis Set (FAS) using a Modified Intent to Treat population.
Measure: Number; unit: percentage of subjects
Arm/Group | NAFT-600 | Placebo
Number analyzed (Participants) | 382 | 179
percentage of subjects
  Mycological Cure | 65.4 | 14.0
  Effective Treatment | 54.2 | 6.1

ADVERSE EVENTS:
Time Frame: Adverse events were collected up to Week 6.
Arm/Group | NAFT-600 | Placebo
Serious Adverse Events (participants affected / at risk) | 2/571 | 2/284
Other Adverse Events (participants affected / at risk) | 13/571 | 2/284
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NAFT-600 (N=571) | Placebo (N=284)
Skull Fractured Base (Injury, poisoning and procedural complications) | 1 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Abscess (Infections and infestations) | 0 | 1
Respiratory Tract Infection (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NAFT-600 (N=571) | Placebo (N=284)
Headache (Nervous system disorders) | 13 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and Principal Investigator agreed not to individually publish or assist other person or entity with any articles, papers, and/or make presentations, speeches referring to the protocol, clinical trial data, the study, or the study drug or any data, results, materials, or information generated or obtained by the Institution or the Principal Investigator without the prior written consent of Merz, which consent may be withheld in the sole discretion of Merz.